CLINICAL TRIAL: NCT03477643
Title: Retrospective Viability Study of the PETHEMA-POMCIDEX Clinical Practice Guidelines for the Treatment of Patients With Relapsed and Refractory Multiple Myeloma (RRMM)
Status: Completed | Type: Observational
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: GEM-POMCIDEX
Record Dates: First submitted 2018-03-13; First posted 2018-03-26 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Relapsed and Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Refractory Multiple Myeloma: Patients with relapsed and refractory multiple myeloma who have received treatment with pomalidomide, cyclophosphamide, and dexamethasone following the GEM-PETHEMA clinical practice guidelines between 01/01/2015 to 01/04/2018

SUMMARY:
Multiple myeloma (MM) is a plasma cell neoplasm representing the second most common type of hematologic tumor after lymphomas. The incorporation of novel agents such as bortezomib, lenalidomide, or thalidomide into first-line treatment as well as in relapse settings has led to a significant improvement in survival rates for MM patients, which have doubled in the last 5-7 years (1,2). However, except for a small percentage of patients (10-30%)(3) that may achieve a cure after first-line treatment, in the majority of cases, MM behaves as an incurable disease whose clinical course is characterized by repeated relapses, shorter and shorter periods of remission, and by becoming refractory to succesive treatments (bortezomib or lenalidomide). In this situation, survival is generally less than 9 months, which underscores the need to develop new drugs for MM patients Pomalidomide, a third-generation immunomodulatory drug (IMiD), has demonstrated efficacy in patients with relapsed and refractory MM, with an overall response rate that fluctuates between 30-60% depending on whether it is administered in combination with low-dose dexamethasone or in association with treatment with a cytostatic agent such as cyclophosphamide.

In clinical trial CC-4047-MM-003, treatment with pomalidomide and low-dose dexamethasone in patients with relapsed and refractory MM or those intolerant to bortezomib or lenalidomide was a successful rescue treatment in 30% of patients with a median progression-free survival of 4 months. The association of cyclophosphamide at dose of 400mg/day on days 1, 8, and 15 of each cycle is able to increase the overall response rate from 39% for combination pomalidomide-dexamethasone to up to 65% for the triple regimen (pomalidomide, cyclophosphamide, dexamethasone - POMCIDEX), as well as the median PFS from 4.4 mo. to 9.2 mo. respectively. As well, the tolerance and safety profiles of the triple combination pomalidomide, cyclophosphamide, and dexamethasone were acceptable.

The association of bortezomib with pomalidomide-dexamethasone also increases the overall response rate (85%) and prolongs PFS (10.7 months).

The BiRD study (lenalidomide, dexamethasone, and clarithromycin) suggests that clarithromycin intensifies the effect of corticosteroids, increasing their anti-myeloma effect . A study evaluating the combination of clarithromycin with pomalidomide and low-dose dexamethasone in RRMM patients showed an overall response rate of 57% and clinical benefit rate (considered equal or superior to minor response) of 66%.

Since July 2014, pomalidomide (Imnovid®) in combination with dexamethasone has been approved for the treatment of adult patients with relapsed and refractory MM who have received at least two prior lines of therapy (including bortezomib and lenalidomide) and who have shown progressive disease to the last line of treatment.

In Spain in January of 2015, and in the Spanish Myeloma Group (GEM) context, we implemented clinical practice guidelines for the treatment of RRMM patients who are candidates for pomalidomide treatment with a triple therapy combination pomalidomide + cyclophosphamide + low-dose dexamethasone (POMCIDEX) (Appendix 1). The goal of the clinical practice guidelines was to increase the overall response rate, quality of response, and progression-free survival in patients treated with POMCIDEX. In patients with suboptimal response (defined as stable disease in the first 3 cycles, or inferior to partial response after six cycles according to International Myeloma Working Group Uniform Response Criteria [7]), clarithromycin can be added to their treatment at a dose of 500mg/12hrs on days 1-28 of each cycle. Treatment can be administered until disease progression, unacceptable toxicity, or based on patient decision.

Keeping in mind the time that has passed since the approval of pomalidomide for use in Spain and the publication of the clinical practice guidelines, we believe it is now time for a retrospective evaluation of the results of the therapeutic guidelines for Spanish MM patients and to review the viability of the recommendations contained in the guidelines with respect to compliance with the same, and effectiveness of the planned course of treatment. Once the viability of the proposed therapy regimen has been evaluated, other analyses for the purpose of studying the clinical results of treatment can be carried out as a separate analysis.

The therapeutic paradigm for MM is rapidly changing due to the availability of new drugs for the treatment of patients with refractory or relapsed disease, making clinical decisions more challenging. For this reason, the availability of data obtained from real-life settings, outside of clinical trials, is essential in order to choose the appropriate treatment for each patient

DETAILED DESCRIPTION:
This is a national, multicentre, observational, retrospective, open-label, non-randomized, non-interventional study to evaluate the degree of compliance at PETHEMA centres in Spain with the clinical practice guidelines proposed by the Spanish Myeloma Group for the treatment of relapsed and refractory MM with POMCIDEX.

In this study, all patients will be included retrospectively who met the inclusion criteria for the GEM clinical practice guidelines and who were treated with POMCIDEX. The period of retrospective data collection will be from 01/01/2015 to 01/04/2018.

The period of data collection for the study includes a maximum period of three months to allow each centre to collect the necessary clinical and demographic data for each patient in order to fulfill the different study objectives. Patient data will be anonymized and recorded in the electronic Case Report Form (eCRF) using the RedCap platform. Afterward, data cleansing and verification will be carried out on all data recorded by the study investigators. This procedure will be carried out in the six months after database lock.

Once the process of recording and verification of patient data is complete, extraction and statistical analysis of the data will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with POMCIDEX during the period 01/01/2015 and 01/04/2018 in accordance with the PETHEMA clinical practice guidelines. The inclusion criteria in the guidelines are those specified in the clinical practice guidelines

Exclusion Criteria:

* Patients who have not been treated according to the clinical practice guidelines during the specified period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with POMCIDEX during the period 01/01/2015 and 01/04/2018 in accordance with the PETHEMA clinical practice guidelines. The inclusion criteria in the guidelines are those specified in the clinical practice guidelines
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Level of compliance at PETHEMA centres in Spain with the clinical practice guidelines proposed by the Spanish Myeloma Group for the treatment of relapsed and refractory MM with POMCIDEX. | 3 months
  To evaluate the viability of the therapeutic guidelines, measured in terms of compliance and the effectiveness of the treatment planned.

CONTACTS AND LOCATIONS:
Locations (27):
- Spain (27):
  - Hospital de Sant Joan de Déu, Barcelona
  - Hospital Donostia-Donostia Ospitalea, Donostia / San Sebastian
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital General San Jorge - Huesca, Huesca
  - Hospital de Jaén, Jaén
  - Hospital Lucus Augusti, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital Del Tajo, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Complejo Hospitalario de Especialidades Virgen de La Victoria, Málaga
  - Hospital Universitario Virgen de La Arrixaca, Murcia
  - Hospital Central de Asturias, Oviedo
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital El Bierzo, Ponferrada
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Mutua Terrassa, Terrassa
  - Complejo Hospitalario de Toledo, Toledo
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Universitario Dr. Peset Aleixandre, Valencia
  - Hospital Universitario La Fe, Valencia
  - HOSPITAL CLíNICO UNIVERSITARIO DE VALLADOLID, Valladolid
  - Hospital Txagorritxu, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://fundacionpethema.es